CLINICAL TRIAL: NCT03974061
Title: Brief Acceptance and Commitment Therapy for HIV-infected At-risk Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-278
Record Dates: First submitted 2019-05-10; First posted 2019-06-04 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Treatment
Keywords: Brief Acceptance and Commitment Therapy; HIV; Alcohol; Randomized Controlled Trial
MeSH Terms: interventions — Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (stratified by gender and interventionist) to a treatment condition (brief acceptance and commitment therapy or a brief alcohol intervention) and an interventionist.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to which intervention is hypothesized to be superior and produce the intended effects. Outcome assessors will be blinded to which intervention participants received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Acceptance and Commitment Therapy (Experimental): Participants randomized to the Acceptance and Commitment Therapy (ACT) arm will receive one, 1-hour intervention session followed by five weekly 30-45 minute intervention sessions delivered via telephone.
  Interventions: Behavioral: Brief Acceptance and Commitment Therapy
- Brief Alcohol Intervention (Active Comparator): Participants randomized to the Brief Alcohol Intervention (BI) will receive the following telephone-based sessions over the duration of six weeks: a 30-45 minute session of a brief alcohol intervention, a 5-10 minute booster call, a reminder phone call for the next intervention session, a 30-45 minute intervention session, a 5-10 minute booster, and a reminder phone call for the post-treatment appointment.
  Interventions: Behavioral: Brief Alcohol Intervention

INTERVENTIONS:
Behavioral: Brief Acceptance and Commitment Therapy — Acceptance and Commitment Therapy utilizes mindfulness skills and values-guided behavioral action plans to decrease experiential avoidance and impact a broad array of psychological symptoms.
  Other Names: Brief ACT
  Arms: Brief Acceptance and Commitment Therapy
Behavioral: Brief Alcohol Intervention — The Brief Alcohol Intervention is a standard intervention that will be adapted for men and women living with HIV. The intervention will be matched in frequency and length to the brief ACT intervention.
  Other Names: BI
  Arms: Brief Alcohol Intervention

SUMMARY:
Alcohol consumption at hazardous levels is associated with negative consequences on nearly every step of the HIV care continuum. It is a critical factor in HIV treatment that, if unaddressed, significantly contributes to onward transmission and poor treatment outcomes. Alcohol interventions for people living with HIV (PLWH) in the United States (US) have shown mixed results, and no alcohol intervention for PLHW has shown long-term reductions in heavy drinking or a significant impact on HIV-related outcomes. One hypothesized reason for this limited success is the failure of these interventions to address the multiple overlapping problems (e.g., comorbid mental health conditions, behavioral health needs) of PLWH who are hazardous drinkers. Innovative alcohol intervention strategies that can have an impact on these multiple behavioral health needs, in a format that can be feasibly delivered in the context of HIV care, are needed. Brief Acceptance and Commitment Therapy (ACT) is a promising intervention for HIV-infected hazardous drinkers. ACT is a transdiagnostic treatment that uses mindfulness skills and values-guided behavioral action plans to impact a broad array of psychological symptoms. ACT has shown efficacy for treatment of anxiety, depression, chronic pain, and substance use, making it a promising approach for hazardous drinkers. The overall objective of this application is to adapt an existing brief ACT intervention developed for smoking cessation, and pilot test its feasibility and acceptability for PLWH who are hazardous drinkers. We hypothesize that the resulting intervention will be preliminarily associated with decreased alcohol use, improved ART adherence, decreased symptoms of depression, anxiety, and drug use, and increased acceptance-a known mechanism of change in ACT.

DETAILED DESCRIPTION:
Alcohol use is a major problem in HIV care. Sixty-six percent of people living with HIV (PLWH) report using alcohol in the previous year, 8-20% report drinking at hazardous or heavy levels, and 30% report current binge drinking (>5 drinks in an occasion in the past 30 days). PLWH who are hazardous drinkers, compared to those who abstain, experience a significant increased risk for: taking ART medications off schedule, suboptimal adherence to ART, and engaging in sexual risk behavior. Hazardous alcohol consumption has been found to affect every stage of the HIV care continuum, from diagnosis, to linkage to care, to retention, and viral suppression, making it a critical factor in HIV treatment that, if unaddressed, may significantly contribute to onward transmission.

Behavioral interventions for HIV-infected drinkers have provided limited evidence of benefit. HIV-prevention interventions do not typically address alcohol use, and it is often overlooked in HIV care. While there have been several clinical trials of alcohol interventions for PLWH in the US, these trials have shown mixed results for reducing alcohol use and improving HIV-related outcomes. No alcohol intervention for PLHW has shown long-term reductions in heavy drinking or a significant impact on HIV-related outcomes. One hypothesized reason for this limited success is that PLWH who are at-risk drinkers are also likely to have multiple overlapping problems. It is estimated that 38% of PLWH meet criteria for both a substance use and another psychiatric disorder and also have a myriad of behavioral health needs (e.g., treatment adherence, condom use), any one of which would benefit from intervention. In order to adequately address these issues, PLWH require innovative alcohol intervention strategies that can also have an impact on other behavioral and mental health needs, in a format that can be feasibly delivered in the context of HIV care.

Brief acceptance and commitment therapy (ACT) is a promising intervention for HIV-infected drinkers. ACT is a transdiagnostic treatment that targets experiential avoidance (repeated attempts to eliminate or avoid difficult thoughts/feelings) as an underlying factor common to mental and behavioral health problems. Mindfulness skills and values-guided behavioral action plans are used to decrease experiential avoidance and impact a broad array of psychological symptoms. ACT has shown efficacy for treatment of anxiety depression, and chronic pain, making it a promising approach for HIV-infected hazardous drinkers. A recently published meta-analysis also indicates that ACT is efficacious for smoking, opiate use, methamphetamine use, and polydrug abuse, showing a small to medium effect size compared to active treatment controls (e.g., Cognitive Behavioral Therapy (CBT), pharmacotherapy). ACT's unique focus on skills that increase the ability to experience and accept, rather than change and control, urges and cravings related to substance use is different from more traditional forms of addiction treatment such as CBT. Indeed, a pilot RCT of a brief, telephone-delivered ACT intervention for smoking cessation had quit rates more than double that of traditional CBT for smokers with comorbid depression. However, ACT has not been studied as an intervention for hazardous drinkers.

The overall objective of this study is to adapt an existing brief ACT intervention and pilot test its feasibility, acceptability, and preliminary efficacy for PLWH who are hazardous drinkers. We hypothesize that the resulting intervention will have a significant effect on biological and self-reported measures of alcohol use and ART adherence. Secondary analyses will also examine changes in acceptance-a known mechanism of change in ACT -symptoms of depression and anxiety, and drug use, which we expect to differ by treatment group. The specific aims are as follows:

Aim 1: Adapt an existing brief ACT intervention for HIV-infected at-risk drinkers (ACT). We will accomplish this aim by: Modifying an existing 5-session, telephone-delivered ACT intervention for smoking cessation using a theoretical framework that has been previously used to systematically adapt evidence-based HIV interventions. We will conduct iterative multidisciplinary team meetings, focus group discussions with HIV clinic patients (N = 15-20), and qualitative interviews with HIV clinic providers (N = 5-10) to inform the adaptation process, get feedback on intervention content, and develop a new treatment manual.

Aim 2: Conduct a pilot superiority trial of ACT compared to a brief alcohol intervention. We will accomplish this aim by: Randomly assigning N = 74 HIV-infected hazardous drinkers (50% women) to the intervention developed in Aim 1 (n = 30) or a brief alcohol intervention previously developed for PLWH that is nearly equivalent in number and length of sessions. We will assess feasibility, acceptability, and primary trial outcomes of alcohol use and ART adherence immediately post-treatment and again at 3 and 6-months post-randomization. Secondary outcomes of changes in acceptance, symptoms of depression, symptoms of anxiety, and drug use will be assessed at all time points.

The proposed research will provide essential pilot data for an R01 application to conduct a full-scale RCT to determine the efficacy of ACT compared with the current evidence-based treatment for PLWH. If successful, this intervention will have broad implications for implementation in HIV and other integrated care settings.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age,
2. HIV-positive,
3. currently prescribed ART medication,
4. score of ≥4 (men) or ≥3 (women) on the AUDIT-C.

Exclusion Criteria:

1. Experiencing acute illness or declining health status when it is determined by a treatment provider that research participation is contraindicated,
2. unable to understand spoken English,
3. does not own a cell phone,
4. a score of 12 on the AUDIT-C, indicating high risk for a severe alcohol use disorder,
5. a score of ≥20 on the PHQ-9 indicating severe depressive symptoms,
6. a score of ≥15 on the GAD-7, indicating severe symptoms of anxiety,
7. experiencing active psychosis as judged by research staff via scores on the BSI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Change in alcohol consumption from baseline to 7-weeks post-treatment | Change in alcohol consumption will be measured via the TLFB from baseline to end of treatment at 7-weeks.
  Alcohol consumption will be measured by retrospective self-report via the Time Line Follow Back (TLFB) interview method which yields the following: number of drinks per drinking day, number of heavy drinking (>3 for women; >4 for men) episodes, and number of drinking days over the last 42-day period.
Change in alcohol consumption from 7-weeks post-treatment to 3-months post-baseline | Change in alcohol consumption will be measured via the TLFB from 7-weeks post-treatment to 3-months post-baseline.
  Alcohol consumption will be measured by retrospective self-report via the Time Line Follow Back (TLFB) interview method which yields the following: number of drinks per drinking day, number of heavy drinking (>3 for women; >4 for men) episodes, and number of drinking days over the last 42-day period.
Change in alcohol consumption from 3-months post-baseline to 6-months post-baseline | Change in alcohol consumption will be measured via the TLFB from 3-months post-baseline to 6-months post-baseline.
  Alcohol consumption will be measured by retrospective self-report via the Time Line Follow Back (TLFB) interview method which yields the following: number of drinks per drinking day, number of heavy drinking (>3 for women; >4 for men) episodes, and number of drinking days over the last 42-day period.
Change in alcohol consumption from baseline to 6-months post-baseline | Change in alcohol consumption will be measured via PEth from baseline to 6-months post-baseline.
  Alcohol use will also be assessed using the biomarker phosphatidylethanol (PEth). PEth is an abnormal phospholipid formed only in the presence of alcohol with an estimated half-life of 4-12 days and can be measured from dried blood spots.
Change in ART adherence from baseline to 7-weeks post-treatment | Change in ART adherence will be measured via VAS from baseline to end of treatment at 7-weeks.
  Adherence will be measured by self-report via the validated visual analog scale (VAS) to identify participants will optimal (>95%) versus suboptimal (<95%) adherence. The VAS asks participants to point to the place on a line ranging from 0-100% that best represents how much of their ART medication that they have taken in the last month.
Change in ART adherence from 7-weeks post-treatment to 3-months post-baseline | Change in ART adherence will be measured via VAS from 7-weeks post-treatment to 3-months post-baseline.
  Adherence will be measured by self-report via the validated visual analog scale (VAS) to identify participants will optimal (>95%) versus suboptimal (<95%) adherence. The VAS asks participants to point to the place on a line ranging from 0-100% that best represents how much of their ART medication that they have taken in the last month.
Change in ART adherence from 3-months post-baseline to 6-months post-baseline | Change in ART adherence will be measured via VAS from 3-months post-baseline to 6-months post-baseline.
  Adherence will be measured by self-report via the validated visual analog scale (VAS) to identify participants will optimal (>95%) versus suboptimal (<95%) adherence. The VAS asks participants to point to the place on a line ranging from 0-100% that best represents how much of their ART medication that they have taken in the last month.
Change in ART adherence from baseline to 6-months post-baseline | Change in ART adherence will be measured via ARV levels in hair from baseline to 6-months post-baseline.
  Adherence will also be measured via ARV levels in hair. Hair concentrations of ARVs have been shown to be the strongest independent predictor of virological success in prospective cohorts of HIV-infected patients.

SECONDARY OUTCOMES:
Acceptance | Acceptance will be measured at baseline, 7-weeks post-baseline, and 3 and 6-month follow-ups.
  Acceptance will be measured using the total score obtained via the self-report Brief Experiential Avoidance Questionnaire (BEAQ). The BEAQ is a 15-item measures that assesses six domains of experiential avoidance: behavioral avoidance, distress aversion, procrastination, distraction, repression/denial and distress endurance.
Symptoms of Depression | Symptoms of depression will be measured at baseline, 7-weeks post-baseline, and 3 and 6-month follow-ups.
  Symptoms of depression will be measured using the total score obtained via the self-report Patient Health Questionnaire (PHQ)-9. The PHQ-9 is a 10-item standardized measure of depression severity.
Symptoms of Anxiety | Symptoms of anxiety will be measured at baseline, 7-weeks post-baseline, 3 and 6-month follow-ups.
  Symptoms of anxiety will be measured using the total score obtained via the self-report Generalized Anxiety Disorder 7-item (GAD-7). The GAD-7 is a 7-item standardized measure of anxiety severity.
Substance Use | Substance use will be measured at baseline, 7-weeks post-baseline, and 3 and 6-month follow-ups
  Substance use will be measured by retrospective self-report via the Time Line Follow Back (TLFB) interview method which yields the number of days non-prescription drugs were used.

OTHER OUTCOMES:
Chronic Pain | Pain will be measured at baseline, 7-weeks post-baseline, 3 and 6-month follow-ups.
  Pain will be measured using the total score obtained via the self-report brief Graded Chronic Pain Scale (GCPS-PCS). The GCPS-CPS is a 3-item measure that yields both continuous and categorical outcomes of pain.
HIV Medication Adherence Self-Efficacy | HIV Medication Adherence Self-Efficacy will be measured at baseline, 7-weeks post-baseline, 3 and 6-month follow-ups.
  HIV Medication Adherence Self-Efficacy will be measured using the total score obtained via the self-report HIV Treatment Adherence Self-Efficacy Scale (HIV-ASES). The HIV-ASES is a 12-item measure of one's confidence in their ability to adhere to a treatment plan.
Alcohol-Related Problems | Alcohol-related problems will be measured at baseline, 7-weeks post-baseline, 3 and 6-month follow-ups.
  Alcohol-related problems will be measured using the total score obtained from the Short Inventory of Problems (SIP-2L). The SIP-2L is a 15-item measure that assesses negative consequences of alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Woolf-King, PhD, Principal Investigator — Syracuse University; Stephen A Maisto, PhD, Principal Investigator — Syracuse University
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed pilot randomized clinical trail (RCT) will include data from approximately 74 HIV-infected hazardous drinkers recruited from a single HIV clinic. The final dataset will include self-reported demographic and behavioral data related to substance use, HIV medication adherence, and general mental health functioning as well as laboratory data from dried blood spots and hair analysis. We will be collecting identifying information in a separate database to track participants for followup appointments. Even though the final computerized dataset will be stripped of all personal identifiers, given the small sample of the study, and the sole recruitment source, there remains a possibility of deductive disclosure of research participants with unusual characteristics. We will thus make the data and associated documentation available to users only via a signed data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing will be available upon publication of the main study findings.
Access Criteria: We will make the data and associated documentation available to users only via a signed data-sharing agreement that stipulates a commitment to: (1) only use the data for research purposes and not to identify any individual participants, (2) securely storing the data via password-protected databases and secure servers, and (3) destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Woolf-King SE, Dalton MR, Firkey M, Sheinfil A, Bucci V, Estrada B, Ramos J, Hahn JA, Bricker J, Gump B, Bendinskas KG, Maisto SA. A Randomized Feasibility/Acceptability Trial of Acceptance and Commitment Therapy for People with HIV Who Drink at Unhealthy Levels. AIDS Behav. 2025 Dec 29. doi: 10.1007/s10461-025-04990-7. Online ahead of print. PMID 41460282

DOCUMENTS (1):
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03974061/ICF_001.pdf